CLINICAL TRIAL: NCT05101889
Title: Benefits of Immunonutrition in Patients With Head and Neck Cancer Receiving Chemoradiation: A Phase II Randomized, Double-blind Study
Brief Title: Benefits of Immunonutrition in Patients With Head and Neck Cancer Receiving Chemoradiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Arunee Dechaphunkul, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC.56-036-13-1-1
Record Dates: First submitted 2021-09-29; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Oral Mucositis
Keywords: head and neck cancer; nasopharyngeal cancer; immunonutrition; concurrent chemoradiation; survival
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Nasopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: phase II randomized, double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition (Experimental): Oral immunomodulating formula (Oral Impact®, Nestle) One sachet of Oral Impact® consisted of 74 g of powder providing 303 kilocalories.
  Three ready-to-drink bottles contained 303 kilocalories/bottle per day, starting 5 days before each chemotherapy session.
  Interventions: Dietary Supplement: Oral Impact®
- Control (Active Comparator): An isocaloric isonitrogenous standard enteral nutrition formula. Three ready-to-drink bottles contained 303 kilocalories/bottle per day, starting 5 days before each chemotherapy session.
  Interventions: Dietary Supplement: Oral Impact®

INTERVENTIONS:
Dietary Supplement: Oral Impact® — 3 ready-to-drink bottles/day
  Other Names: Blendera®

SUMMARY:
This study evaluated the benefits of immunonutrition regarding the prevention of severe mucositis. Patients with head and neck cancer (HNC) undergoing definitive concurrent chemoradiation including 3-week cycles of cisplatin were enrolled in this double-blind phase II study. Patients were randomly assigned to receive an immunonutrition containing omega-3-fatty acids, arginine, dietary nucleotides, and soluble fiber or an isocaloric isonitrogenous control. All patients received the assigned product 5 days before each chemotherapy session. The proportion of patients with severe mucositis was compared between the immunonutrition and control groups.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-65 years
* histological confirmation of stage II-IVb non-metastatic HNC according to the seventh edition of the American Joint Committee on Cancer Staging System (AJCC 2010)
* receipt of definitive CCRT
* Eastern Cooperative Oncology Group performance status of 0-1
* creatinine clearance ≥ 60 mL/min/1.73 m2 calculated by the Cockcroft-Gault formula
* absence of mucositis
* able to tolerate oral feeding

Exclusion Criteria:

* receipt of curative surgery for HNC
* allergies to any component of the immunonutrition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Severe oral mucositis graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 criteria | 6 weeks after initiation of concurrent chemoradiation (CCRT)
  Proportion of severe oral mucositis between two groups

SECONDARY OUTCOMES:
Other treatment-related toxicities graded according to the NCI CTCAE version 4.03 criteria | through study completion, an average of 6 weeks
  Proportion of patients with other treatment-related toxicities between two groups
body weight in kilograms | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean changes of body weight between two groups
serum albumin in grams per deciliter (g/dL) | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean serum albumin between two groups
hemoglobin in grams per deciliter (g/dL) | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean hemoglobin between two groups
C-reactive protein (CRP) in milligrams per liter (mg/L) | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean CRP between two groups
neutrophil-to-lymphocyte ratio (NLR) | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean NLR between two groups
platelet-to-lymphocyte ratio (PLR) | 6 weeks after initiation of CCRT and 1 month after CCRT completion
  mean PLR between two groups
actual dose of radiation in centigrays (cGy) | through study completion, an average of 6 weeks
  mean actual dose of radiation between two groups
cumulative dose of cisplatin in milligrams per square meter (mg/m2) | through study completion, an average of 6 weeks
  mean cumulative dose of cisplatin between two groups
progression-free survival (PFS) | at 3 years
  compare PFS between two groups
overall survival (OS) | at 3 years
  compare OS between two groups

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dechaphunkul T, Arundon T, Raungkhajon P, Jiratrachu R, Geater SL, Dechaphunkul A. Benefits of immunonutrition in patients with head and neck cancer receiving chemoradiation: A phase II randomized, double-blind study. Clin Nutr. 2022 Feb;41(2):433-440. doi: 10.1016/j.clnu.2021.12.035. Epub 2021 Dec 28. PMID 35007812